CLINICAL TRIAL: NCT00528190
Title: Treatment of Aspergillus Fumigatus in Patients With Cystic Fibrosis: A Randomized, Double-blind, Placebo-Controlled Trial
Brief Title: Treatment of Aspergillus Fumigatus (a Fungal Infection) in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Hospital for Sick Children (Other); Canadian Cystic Fibrosis Foundation (Other); The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2006768
Record Dates: First submitted 2007-09-10; First posted 2007-09-12 (Estimated); Results first posted 2017-03-23 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Aspergillus Fumigatus; randomized controlled clinical trials
MeSH Terms: conditions — Cystic Fibrosis | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itraconazole (Experimental): Itraconazole 5mg/kg/day for 24 weeks
  Interventions: Drug: Itraconazole
- Placebo (Placebo Comparator): Placebo/day for 24 weeks
  Interventions: Drug: Itraconazole

INTERVENTIONS:
Drug: Itraconazole — Oral Itraconazole 5mg/kg/day or identical placebo for 24 weeks
  Other Names: non applicable

SUMMARY:
This clinical trial will attempt to determine whether we can improve clinical outcomes for patients with cystic fibrosis who are infected with a fungus called Aspergillus fumigatus.

DETAILED DESCRIPTION:
The aim of this study is to determine whether antibiotic treatment directed against Aspergillus Fumigatus will be effective at preventing respiratory exacerbations and improving pulmonary function in patients with cystic fibrosis(CF) who are chronically colonized/infected with aspergillus. This aim will be accompanied by means of a randomized, double-blind, placebo-controlled clinical trial incorporating two parallel treatment arms.

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of CF as defined by two or more clinical features of CF and a documented sweat chloride greater than 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease causing mutations
* Patient must be known to be chronically colonized with Aspergillus fumigatus.
* Patients must be clinically stable at randomization, no use of new inhaled, oral or intravenous antibiotics or oral or intravenous corticosteroids during the 14-day period prior to randomization.
* 6 years of age and older
* Patients must weigh at least 20 kg
* Post-menarche females must be using an effective form of contraception.

Exclusion Criteria

* Inability to give informed consent.
* Respiratory culture positive for B.cepacia complex
* Renal function abnormalities-Creatinine greater than 1.5 times upper limit of normal within a 30 day period prior to randomization
* Liver function abnormalities : AST or ALT greater or equal to 2.5 times the upper limit of normal within a 30 day period prior to randomization
* Neutropenia, absolute neutrophil count< or = 1000 within a 3-day period prior to randomization
* History of biliary cirrhosis documented by liver biopsy or imaging.
* History of portal hypertension.
* Investigational drug use within 30 days of randomization date.
* History of alcohol, illicit drug or medication abuse within 1 year of randomization.
* Women who are pregnant, breastfeeding or trying to conceive

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-10; Primary Completion 2010-08 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Aaron, MD, Principal Investigator — OHRI
Locations (2):
- Canada (2):
  - Shawn Aaron, The Ottawa Hospital-General Campus, Ottawa, Ontario
  - Felix Ratjen, The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aaron SD, Vandemheen KL, Freitag A, Pedder L, Cameron W, Lavoie A, Paterson N, Wilcox P, Rabin H, Tullis E, Morrison N, Ratjen F. Treatment of Aspergillus fumigatus in patients with cystic fibrosis: a randomized, placebo-controlled pilot study. PLoS One. 2012;7(4):e36077. doi: 10.1371/journal.pone.0036077. Epub 2012 Apr 30. PMID 22563440

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole: Itraconazole 5mg/kg/day
  Itraconazole: Oral Itraconazole 5mg/kg/day or identical placebo for 24 weeks
Period: Overall Study
Arm/Group | Itraconazole | Placebo
Started | 18 | 17
Completed | 18 | 16
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itraconazole | Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (10.5) | 25.2 (9.1) | 25.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure Will be the Number of Patients Who Experience a Respiratory Exacerbation Requiring Intravenous Antibiotics in the Two Treatment Groups Over the 24 Week Trial Treatment Period.
Description: The Primary outcome measure will be the number of patients who experience a respiratory exacerbation requiring intravenous antibiotics in the two treatment groups over the 24 week trial treatment period.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Itraconazole | Placebo
Number analyzed (Participants) | 18 | 16
Participants | 4 | 5

ADVERSE EVENTS:
Arm/Group | Itraconazole | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/17
Other Adverse Events (participants affected / at risk) | 2/18 | 2/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=18) | Placebo (N=17)
Spontaneous Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole (N=18) | Placebo (N=16)
Increased Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Hemoptysis (Gastrointestinal disorders) | 2 | 1
Hyperglycemia (Endocrine disorders) | 1 | 0
Flu-like Illness (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Conjuctivitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No